CLINICAL TRIAL: NCT00780052
Title: Infusional C-myb Antisense Oligodeoxynucleotide in Advanced Hematological Malignancies
Brief Title: Infusional C-myb ASODN in Advanced Hematologic Malignancies
Acronym: UPCC 04701
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 04701
Record Dates: First submitted 2008-10-24; First posted 2008-10-27 (Estimated); Last update posted 2016-09-26 (Estimated); Status verified 2011-12

CONDITIONS: Hematologic Malignancies
Keywords: Hematologic Malignancies; c-myb; c-myb AS ODN
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Genes, myb

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): c-myb AS ODN as a 24-hour continuous infusion over 7 days
  Interventions: Drug: c-myb AS ODN

INTERVENTIONS:
Drug: c-myb AS ODN — Subjects will be admitted to the hospital to receive c-myb AS ODN as a 24-hour continuous intravenous infusion over 7 days. Dose level is increased with each new subject to determine if there is a MTD.

SUMMARY:
The purpose of this study is to evaluate whether C-myb Antisense (AS) Oligonucleotides (ODNs)is a possible treatment modality for advanced hematologic malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have one of the following: acute myeloid or lymphoid leukemia; or Myeloproliferative disorder(MPD) including Chronic Myelogenous Leukemia (CML); or Myelodysplastic Syndrome (MDS); or Non-Hodgkin's Lymphoma (including CLL); or Multiple Myeloma
* Patients with acute leukemia must meet one of the following conditions:

  *have disease which is refractory to a course of standard induction chemotherapy *have relapsed diseased after documentation of previous clinical remission or *have untreated disease and not be a candidate for conventional first line treatment
* Patients with CML or other MPD must have evidence of accelerated phase or blast crisis
* Patients having clinical features of CML in transformation but who are negative for Philadelphia chromosome may be entered provided there is a prior definable chronic phase
* Patients with Philadelphia chromosome positive CML must have failed treated with Gleevec (Imatinib) in order to be eligible for study
* Patients with myelodysplastic syndrome (MDS) must have > 5% blasts in the peripheral blood or bone marrow and have at diagnosis as IPSS score of >= 1
* Patients with CLL must have relapsed or refractory disease after at least three courses of conventional therapy and have been determined to no longer be a candidate for conventional therapy
* Patients with non-Hodgkin's lymphoma (other than CLL) must have relapsed or refractory disease after at least two courses of chemotherapy and have been determined not to be a candidate for further conventional therapies
* Patients with multiple myeloma must have failed at least 3 prior therapies
* Performance Status 0, 1 or 2
* Serum creatinine < 2.0 mg/dl; serum bilirubin < 2 mg/dl and AST/ALT < 3.0 x upper limit of normal
* PTT within normal range
* Age > 18
* Patients must have an indwelling central venous catheter

Exclusion Criteria:

* Significant cardiac disease which requires active therapy
* Intercurrent organ damage or medical problems that will jeopardize outcome of therapy
* Pregnant or lactating females
* Received prior c-myb AS ODN therapy
* Patients with suitable HLA identical sibling donor who are deemed to be appropriate and willing candidates for allogeneic bone marrow transplantation
* Patients requiring anticoagulation with unfractionated heparin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2002-09; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicities and maximum tolerated dose and maximum tolerated duration of c-myb AS ODN | At study completion

CONTACTS AND LOCATIONS:
Overall Officials: Selina Luger, MD, Principal Investigator — University of Pennsylvania Abramson Cancer Center
Locations (1):
- University of Pennsylvania Abramson Cancer Center, Philadelphia, Pennsylvania, United States